CLINICAL TRIAL: NCT06324695
Title: DEVISE - Development and Evaluation of an Online Intervention to Reduce Self-stigma in People With Visible Chronic Skin Diseases: a Randomized Controlled Trial
Brief Title: Development and EValuation of an Online Intervention to Reduce Self-Stigma in People With Visible Chronic Skin disEases
Acronym: DEVISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01GY2105
Record Dates: First submitted 2023-10-04; First posted 2024-03-22 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis; Alopecia Areata; Hidradenitis Suppurativa; Vitiligo; Atopic Dermatitis
Keywords: Self-compassion; Self-stigma; Cognitive-behavioral therapy; Internet-based intervention; Visible chronic skin disease
MeSH Terms: conditions — Psoriasis; Alopecia Areata; Hidradenitis Suppurativa; Vitiligo; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HautKompass intervention (Experimental): Participants in the intervention group will attend the self-guided 8-session online psychosocial intervention HautKompass.
  Interventions: Behavioral: HautKompass
- Waiting list (No Intervention): Participants in the control group will not attend any psychosocial intervention during the course of the RCT (waiting list). They will be offered the opportunity to attend the HautKompass program after the follow-up phase.

INTERVENTIONS:
Behavioral: HautKompass — The HautKompass program is a structured self-guided online psychosocial intervention designed to reduce self-stigma in people with visible chronic skin diseases. It combines educational content and practical exercises based on cognitive-behavioral therapy (CBT), namely cognitive restructuring of negative automatic thoughts and cultivating self-compassionate thinking and behavior. The program consists of eight skin-generic modules (on average, 15-20 minutes per module, one module per week).
  Arms: HautKompass intervention

SUMMARY:
This project aims to develop and evaluate an online intervention to prevent and/or reduce self-stigma in German patients with visible chronic skin diseases. Evaluation of the intervention with regard to effectiveness and feasibility will follow an open-label randomized controlled design with 550 patients in total. The results of the program are expected to provide new insights and markedly extended knowledge on the mechanisms of self-stigma in chronic skin conditions. The new online intervention can be used in routine care, aiming for better patient care in practice and, ultimately decreased extent of self-stigma, increased quality of life of patients, and decreased rates of depression, anxiety, and suicide ideation.

DETAILED DESCRIPTION:
Background: Approximately 10 million people in Germany suffer from a chronic skin disease. Besides physical symptoms, the psychosocial burden for patients is high. A specific problem is stigmatization, which is still very burdensome for people with skin diseases. As a consequence of experienced discrimination, patients tend to accept and incorporate social prejudices, which impair self-esteem and self-efficacy, enhance isolation, and maintain a negatively self-reinforcing cycle. The World Health Organization has explicitly pointed out the importance of reducing stigma. While recent interventions for reducing external stigma in skin diseases have been developed and positively evaluated, evidence-based interventions on self-stigma in skin diseases are still lacking.

Objective: This project aims to develop and evaluate the effectiveness of an online intervention for patients with psoriasis, atopic dermatitis, hidradenitis suppurativa, alopecia areata, and vitiligo, to prevent and/or reduce self-stigma.

Methods: The evaluation of the online program will follow a randomized controlled design. 550 patients will be recruited through several participating centers across Germany and allocated to the intervention or the control group in a ratio of 1:1, with an equal distribution by diagnosis. Participants in the intervention group will attend a self-guided online program consisting of eight skin-generic modules (on average, 15-20 minutes per module, one module per week), combining educational content and cognitive-behavioral therapy-based exercises (e.g., cognitive restructuring of negative automatic thoughts; cultivating self-compassionate thinking and behavior). Participants in the control group will not attend an alternative program (waiting list) and will be offered the opportunity to attend the program after the follow-up phase. The primary outcome will be a reduction in self-stigma; the secondary outcome will be an improvement in psychosocial health, namely quality of life, depression, anxiety, and suicide ideation. These outcomes will be assessed by standardized patient-reported outcome measures at three time points: baseline (t0), immediately after the intervention (t1), and 6-month follow-up (t2).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis, atopic dermatitis, hidradenitis suppurativa, alopecia areata, or vitiligo;
* Age ≥ 18 years;
* Sufficient language skills (German) to follow the instructions and content of the intervention;
* Access to a desktop/ laptop with internet connection;
* Having signed an Informed Consent Form (ICF).

Exclusion Criteria:

* Age < 18 years;
* Lack of informed consent (ICF);
* Patients that were treated in the last 12 months by a psychologist, psychotherapist, or psychiatrist for major depression, schizophrenia or other psychotic disorder, major bipolar disorder, major anxiety or obsessive-compulsive disorder, post-traumatic stress disorder, or major personality disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to post-intervention and follow-up in self-stigma | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the Weight Bias Internalization Scale (WBIS) - adapted for skin disease. The scale includes 10 items with a Likert-type response scale ranging from 1 to 7 and provides a total sum score ranging from 10 to 70, with higher scores indicating higher internalization of stigma and biases associated with own skin disease.

SECONDARY OUTCOMES:
Changes from baseline to post-intervention and follow-up in generic quality of life | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the EUROHIS-QOL 8-item index. The instrument includes 8 items assessing overall QOL, general health, energy, daily life activities, esteem, relationships, finances, and home environment, to be scored on a 5-point Likert scale. A total score is generated, with higher scores indicating better quality of life.
Changes from baseline to post-intervention and follow-up in skin-generic quality of life | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the Dermatology Life Quality Index (DLQI), which includes 10 items, to be answered on a 4-point Likert scale ranging from 0 ("not at all"/ "not relevant") to 3 ("very much"). A total sum score ranging from 0 to 30 is computed, with higher scores indicating larger impairments. According to the Hongbo classification, DLQI scores > 10 are considered as large or extremely large impairments on patients' life.
Changes from baseline to post-intervention and follow-up in depression | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the nine-item Patient Health Questionnaire (PHQ-9), which is a validated screening measure for diagnosing and monitoring depression. The response scale ranges from 0 ("not at all") to 3 ("nearly every day"); the sum score ranges from 0 to 27 and a cut-off point ≥ 10 has showed maximized sensitivity and specificity to detect major depression.
Changes from baseline to post-intervention and follow-up in anxiety | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the General Anxiety Disorder (GAD-7), which is a brief validated instrument to screen for anxiety disorders. It comprises seven items that represent core anxiety symptoms. The response scale ranges from 0 ("not at all") to 3 ("nearly every day"); the 7 items can be summed into a total score ranging from 0 to 21, with scores ≥ 10 indicating high likelihood of clinical anxiety disorders.
Changes from baseline to post-intervention and follow-up in suicidal ideation | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with Paykel's Suicidal Feelings in the General Population Questionnaire, which is one of the most widely used measures of suicidal ideation in different populations, including medical settings. It comprises 5 questions about life-weariness, death wishes, and suicidal thoughts, plans and attempts, to be answered in a yes/no response scale. A "yes"-response to questions 3 to 5 indicates the presence of suicidal ideation.
Feasibility of the HautKompass online program | continuously tracked during intervention
  Measured through general statistics of website utilization (e.g., time spent on each session). Durations of individuals sessions of > 45 minutes are considered not feasible for implementation.
Feasibility of the HautKompass online program - dropouts | continuously tracked during intervention
  Measured through dropout rate.
User satisfaction with the HautKompass online program | Immediately post-intervention (t1)
  Evaluated with the Client Satisfaction Questionnaire Adapted to Internet-Based Interventions (CSQ-I), which includes 8 questions on a Likert scale of 1 to 4, with higher scores indicating greater satisfaction.
Acceptability of the HautKompass online program | Immediately post-intervention (t1)
  Evaluated with an ad hoc questionnaire that comprises 5 questions about the general acceptability of the website. Respondents are asked to answer the questions on a 4-point Likert scale, where higher scores represent higher acceptability.

OTHER OUTCOMES:
Changes from baseline to post-intervention and follow-up in illness identity | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the Inclusion of Illness in the Self (IIS) scale. Respondents indicate in a single item the degree to which their illness is integrated into their self-concept. The higher the IIS score, the greater patients felt they internalized their illness.
Changes from baseline to post-intervention and follow-up in avoidance and acceptance coping | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the subscales avoidance (8 items) and positive rational acceptance (11 items) of the Body Image Coping Strategies Inventory (BICSI). The 19 items are answered in a Likert-type response scale ranging from 0 to 3, and an average score is calculated for each subscale, with higher scores indicating more frequent use of the specific coping strategy.
Changes from baseline to post-intervention and follow-up in generic body image/ appearance concerns | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the Appearance Orientation Subscale of the Multidimensional Body-Self Relations Questionnaire (MBSRQ-AO). This subscale includes 2 items, to be answered on a 5-point Likert scale. The average score for the subscale is computed, with higher scores indicating more appearance concerns.
Changes from baseline to post-intervention and follow-up in cutaneous body image | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the Cutaneous Body Image Scale (CBIS), which comprises 7 items, to be rated on a response scale from 0 ("not at all") to 9 ("very markedly"). A composite score is derived from the mean ratings of the seven items, where a high score is indicative of greater satisfaction with cutaneous body image: score < 3 = severe dissatisfaction; 3-6 = moderate dissatisfaction; > 6 = mild to no dissatisfaction.
Changes from baseline to post-intervention and follow-up in self-compassion | Baseline (t0), immediately post-intervention (t1), 6-months follow-up (t2)
  Evaluated with the short version of the Self-Compassion Scale (SCS), which includes 12 items, to be answered in a 5-point response scale ranging from 1 ("Almost never") to 5 ("Almost always"). Mean scores can be computed for six subscales - Self-Kindness, Self-Judgment (reversed scoring), Common Humanity, Isolation (reversed scoring), Mindfulness, and Over-identification (reversed scoring), as well as a total self-compassion score that results from the average of the six subscale mean scores, with higher scores indicating higher levels of self-compassion.
Session Feedback | At the end of each session of the program
  Evaluated with an ad hoc questionnaire that comprises 3 questions tapping into whether the session just completed was interesting, easy to understand, and personally helpful. Respondents are asked to answer the questions on a 5-point Likert scale, where higher scores represent greater agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sommer, Priv-Doz.Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (12):
- Germany (12):
  - Deutscher Vitiligo-Bund e.V., Adelsdorf
  - Fachklinik Bad Bentheim, Fachbereich Dermatologie und Allergologie, Bad Bentheim
  - Universitätsklinikum der Ruhr-Universität Bochum (UKRUB), Klinik für Dermatologie, Venerologie und Allergologie, Bochum
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Institut für Versorgungsforschung in der Dermatologie und bei Pflegeberufen (IVDP), Hamburg
  - Deutscher Psoriasis Bund e.V. (DPB), Hamburg
  - Hautarztpraxis Dr. Daniela Kasche, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Klinik für Dermatologie, Venerologie und Allergologie, Psoriasis-Zentrum-Kiel, Kiel
  - Alopecia Areata Deutschland e.V., Krefeld
  - Universitätsmedizin der Johannes-Gutenberg-Universität Mainz, Hautklinik und Poliklinik, Mainz
  - Technische Universität München, Klinik und Poliklinik für Dermatologie und Allergologie am Biederstein, München
  - Universitätsklinikum Münster (UKM), Klinik für Hautkrankheiten - Allgemeine Dermatologie und Venerologie, Münster
  - Dermatologische Spezial- und Schwerpunktpraxis Dr. med. Ralph von Kiedrowski, Selters

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bessell A, Brough V, Clarke A, Harcourt D, Moss TP, Rumsey N. Evaluation of the effectiveness of Face IT, a computer-based psychosocial intervention for disfigurement-related distress. Psychol Health Med. 2012;17(5):565-77. doi: 10.1080/13548506.2011.647701. Epub 2012 Feb 7. PMID 22313169
- [Background] Durso LE, Latner JD. Understanding self-directed stigma: development of the weight bias internalization scale. Obesity (Silver Spring). 2008 Nov;16 Suppl 2:S80-6. doi: 10.1038/oby.2008.448. PMID 18978768
- [Background] Schmidt S, Muhlan H, Power M. The EUROHIS-QOL 8-item index: psychometric results of a cross-cultural field study. Eur J Public Health. 2006 Aug;16(4):420-8. doi: 10.1093/eurpub/cki155. Epub 2005 Sep 1. PMID 16141303
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lowe B, Kroenke K, Herzog W, Grafe K. Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). J Affect Disord. 2004 Jul;81(1):61-6. doi: 10.1016/S0165-0327(03)00198-8. PMID 15183601
- [Background] Paykel ES, Myers JK, Lindenthal JJ, Tanner J. Suicidal feelings in the general population: a prevalence study. Br J Psychiatry. 1974 May;124(0):460-9. doi: 10.1192/bjp.124.5.460. No abstract available. PMID 4836376
- [Background] Cash TF, Santos MT, Williams EF. Coping with body-image threats and challenges: validation of the Body Image Coping Strategies Inventory. J Psychosom Res. 2005 Feb;58(2):190-9. doi: 10.1016/j.jpsychores.2004.07.008. PMID 15820848
- [Background] Vossbeck-Elsebusch AN, Waldorf M, Legenbauer T, Bauer A, Cordes M, Vocks S. German version of the Multidimensional Body-Self Relations Questionnaire - Appearance Scales (MBSRQ-AS): confirmatory factor analysis and validation. Body Image. 2014 Jun;11(3):191-200. doi: 10.1016/j.bodyim.2014.02.002. Epub 2014 Mar 28. PMID 24958652
- [Background] Gupta MA, Gupta AK. Evaluation of cutaneous body image dissatisfaction in the dermatology patient. Clin Dermatol. 2013 Jan-Feb;31(1):72-9. doi: 10.1016/j.clindermatol.2011.11.010. PMID 23245977
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Hilbert A, Baldofski S, Zenger M, Lowe B, Kersting A, Braehler E. Weight bias internalization scale: psychometric properties and population norms. PLoS One. 2014 Jan 29;9(1):e86303. doi: 10.1371/journal.pone.0086303. eCollection 2014. PMID 24489713
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Boss L, Lehr D, Reis D, Vis C, Riper H, Berking M, Ebert DD. Reliability and Validity of Assessing User Satisfaction With Web-Based Health Interventions. J Med Internet Res. 2016 Aug 31;18(8):e234. doi: 10.2196/jmir.5952. PMID 27582341
- [Background] Lara MA, Patino P, Tiburcio M, Navarrete L. Satisfaction and Acceptability Ratings of a Web-Based Self-help Intervention for Depression: Retrospective Cross-sectional Study From a Resource-Limited Country. JMIR Form Res. 2022 Apr 4;6(4):e29566. doi: 10.2196/29566. PMID 35377324
- [Background] Augustin M, Herberger K, Hintzen S, Heigel H, Franzke N, Schafer I. Prevalence of skin lesions and need for treatment in a cohort of 90 880 workers. Br J Dermatol. 2011 Oct;165(4):865-73. doi: 10.1111/j.1365-2133.2011.10436.x. PMID 21623753
- [Background] Dalgard FJ, Gieler U, Tomas-Aragones L, Lien L, Poot F, Jemec GBE, Misery L, Szabo C, Linder D, Sampogna F, Evers AWM, Halvorsen JA, Balieva F, Szepietowski J, Romanov D, Marron SE, Altunay IK, Finlay AY, Salek SS, Kupfer J. The psychological burden of skin diseases: a cross-sectional multicenter study among dermatological out-patients in 13 European countries. J Invest Dermatol. 2015 Apr;135(4):984-991. doi: 10.1038/jid.2014.530. Epub 2014 Dec 18. PMID 25521458
- [Background] Zander N, Sommer R, Schafer I, Reinert R, Kirsten N, Zyriax BC, Maul JT, Augustin M. Epidemiology and dermatological comorbidity of seborrhoeic dermatitis: population-based study in 161 269 employees. Br J Dermatol. 2019 Oct;181(4):743-748. doi: 10.1111/bjd.17826. Epub 2019 Jul 17. PMID 30802934
- [Background] Corrigan PW, Larson JE, Rusch N. Self-stigma and the "why try" effect: impact on life goals and evidence-based practices. World Psychiatry. 2009 Jun;8(2):75-81. doi: 10.1002/j.2051-5545.2009.tb00218.x. PMID 19516923
- [Background] Ali F, Vyas J, Finlay AY. Counting the Burden: Atopic Dermatitis and Health-related Quality of Life. Acta Derm Venereol. 2020 Jun 9;100(12):adv00161. doi: 10.2340/00015555-3511. PMID 32412644
- [Background] Kirsten N, Zander N, Augustin M. Prevalence and cutaneous comorbidities of hidradenitis suppurativa in the German working population. Arch Dermatol Res. 2021 Mar;313(2):95-99. doi: 10.1007/s00403-020-02065-2. Epub 2020 Apr 22. PMID 32322958
- [Background] Radtke MA, Schafer I, Glaeske G, Jacobi A, Augustin M. Prevalence and comorbidities in adults with psoriasis compared to atopic eczema. J Eur Acad Dermatol Venereol. 2017 Jan;31(1):151-157. doi: 10.1111/jdv.13813. Epub 2016 Aug 13. PMID 27521212
- [Background] Titeca G, Goudetsidis L, Francq B, Sampogna F, Gieler U, Tomas-Aragones L, Lien L, Jemec GBE, Misery L, Szabo C, Linder D, Evers AWM, Halvorsen JA, Balieva F, Szepietowski J, Romanov D, Marron SE, Altunay IK, Finlay AY, Salek SS, Kupfer J, Dalgard FJ, Poot F. 'The psychosocial burden of alopecia areata and androgenetica': a cross-sectional multicentre study among dermatological out-patients in 13 European countries. J Eur Acad Dermatol Venereol. 2020 Feb;34(2):406-411. doi: 10.1111/jdv.15927. Epub 2019 Nov 12. PMID 31465592
- [Background] Kage P, Simon JC, Treudler R. Atopic dermatitis and psychosocial comorbidities. J Dtsch Dermatol Ges. 2020 Feb;18(2):93-102. doi: 10.1111/ddg.14029. PMID 32026645
- [Background] Misitzis A, Goldust M, Jafferany M, Lotti T. Psychiatric comorbidities in patients with hidradenitis suppurativa. Dermatol Ther. 2020 Jul;33(4):e13541. doi: 10.1111/dth.13541. Epub 2020 May 22. PMID 32385861
- [Background] Wlodarek K, Glowaczewska A, Matusiak L, Szepietowski JC. Psychosocial burden of Hidradenitis Suppurativa patients' partners. J Eur Acad Dermatol Venereol. 2020 Aug;34(8):1822-1827. doi: 10.1111/jdv.16255. Epub 2020 Mar 10. PMID 32003871
- [Background] Hunt N, McHale S. The psychological impact of alopecia. BMJ. 2005 Oct 22;331(7522):951-3. doi: 10.1136/bmj.331.7522.951. No abstract available. PMID 16239692
- [Background] Rzepecki AK, McLellan BN, Elbuluk N. Beyond Traditional Treatment: The Importance of Psychosocial Therapy in Vitiligo. J Drugs Dermatol. 2018 Jun 1;17(6):688-691. PMID 29879259
- [Background] Ongenae K, Dierckxsens L, Brochez L, van Geel N, Naeyaert JM. Quality of life and stigmatization profile in a cohort of vitiligo patients and effect of the use of camouflage. Dermatology. 2005;210(4):279-85. doi: 10.1159/000084751. PMID 15942213
- [Background] Sommer R, Augustin M, Mrowietz U, Topp J, Schafer I, von Spreckelsen R. [Perception of stigmatization in people with psoriasis-qualitative analysis from the perspective of patients, relatives and healthcare professionals]. Hautarzt. 2019 Jul;70(7):520-526. doi: 10.1007/s00105-019-4411-y. German. PMID 31134287
- [Background] Alpsoy E, Polat M, Yavuz IH, Kartal P, Didar Balci D, Karadag AS, Bilgic A, Arca E, Karaman BF, Emre S, Adisen E, Sendur N, Bilgic O, Cordan Yazici A, Yalcin B, Koca R, Gunduz K, Borlu M, Ergun T, Dursun P, Bilgili SG, Surer Adanir A, Gulekon A, Yagcioglu G, Yilmaz E, Kavuzlu U, Senol Y. Internalized Stigma in Pediatric Psoriasis: A Comparative Multicenter Study. Ann Dermatol. 2020 Jun;32(3):181-188. doi: 10.5021/ad.2020.32.3.181. Epub 2020 Apr 24. PMID 33911736
- [Background] van Beugen S, Maas J, van Laarhoven AI, Galesloot TE, Rinck M, Becker ES, van de Kerkhof PC, van Middendorp H, Evers AW. Implicit stigmatization-related biases in individuals with skin conditions and their significant others. Health Psychol. 2016 Aug;35(8):861-5. doi: 10.1037/hea0000404. PMID 27505208
- [Background] Gonul M, Cemil BC, Ayvaz HH, Cankurtaran E, Ergin C, Gurel MS. Comparison of quality of life in patients with androgenetic alopecia and alopecia areata. An Bras Dermatol. 2018 Sep-Oct;93(5):651-658. doi: 10.1590/abd1806-4841.20186131. PMID 30156613
- [Background] Schmid-Ott G, Kuensebeck HW, Jaeger B, Werfel T, Frahm K, Ruitman J, Kapp A, Lamprecht F. Validity study for the stigmatization experience in atopic dermatitis and psoriatic patients. Acta Derm Venereol. 1999 Nov;79(6):443-7. doi: 10.1080/000155599750009870. PMID 10598757
- [Background] Koumaki D, Efthymiou O, Bozi E, Katoulis AC. Perspectives On Perceived Stigma And Self-Stigma In Patients With Hidradenitis Suppurativa. Clin Cosmet Investig Dermatol. 2019 Oct 16;12:785-790. doi: 10.2147/CCID.S180036. eCollection 2019. PMID 31802927
- [Background] Schmid-Ott G, Kunsebeck HW, Jecht E, Shimshoni R, Lazaroff I, Schallmayer S, Calliess IT, Malewski P, Lamprecht F, Gotz A. Stigmatization experience, coping and sense of coherence in vitiligo patients. J Eur Acad Dermatol Venereol. 2007 Apr;21(4):456-61. doi: 10.1111/j.1468-3083.2006.01897.x. PMID 17373970
- [Background] Wittkowski A, Richards HL, Griffiths CE, Main CJ. The impact of psychological and clinical factors on quality of life in individuals with atopic dermatitis. J Psychosom Res. 2004 Aug;57(2):195-200. doi: 10.1016/S0022-3999(03)00572-5. PMID 15465076
- [Background] Topp J, Andrees V, Weinberger NA, Schafer I, Sommer R, Mrowietz U, Luck-Sikorski C, Augustin M. Strategies to reduce stigma related to visible chronic skin diseases: a systematic review. J Eur Acad Dermatol Venereol. 2019 Nov;33(11):2029-2038. doi: 10.1111/jdv.15734. Epub 2019 Aug 5. PMID 31177601
- [Background] Augustin M, Mrowietz U, Luck-Sikorski C, von Kiedrowski R, Schlette S, Radtke MA, John SM, Zink A, Suthakharan N, Sommer R; German ECHT research group. Translating the WHA resolution in a member state: towards a German programme on 'Destigmatization' for individuals with visible chronic skin diseases. J Eur Acad Dermatol Venereol. 2019 Nov;33(11):2202-2208. doi: 10.1111/jdv.15682. Epub 2019 Jul 8. PMID 31087405
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Barak A, Hen L, Boniel-Nissim M, Shapira N. A comprehensive review and a meta-analysis of the effectiveness of Internet-based psychotherapeutic interventions. Journal of Technology in Human Services 2008; 26(2-4): 109-160.
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Ginsburg IH, Link BG. Feelings of stigmatization in patients with psoriasis. J Am Acad Dermatol. 1989 Jan;20(1):53-63. doi: 10.1016/s0190-9622(89)70007-4. PMID 2913081